CLINICAL TRIAL: NCT03263130
Title: Site and Mechanism(s) of Expiratory Airflow Limitation in COPD, Emphysema and Asthma-COPD Overlap
Status: Recruiting | Type: Observational
Sponsor: Gelb, Arthur F., M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: 1234567
Record Dates: First submitted 2017-08-17; First posted 2017-08-28 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: COPD, Emphysema, Asthma COPD Overlap; Emphysema
Keywords: COPD, Emphysema, Asthma COPD Overlap
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD, Emphysema, Asthma-COPD Overlap: Based on clinical, pathologic, laboratory, physiologic and radiologic differences, patient groups can be described.
  Interventions: Other: As above: diagnosis: COPD, Emphysema, Asthma-COPD Overlap

INTERVENTIONS:
Other: As above: diagnosis: COPD, Emphysema, Asthma-COPD Overlap

SUMMARY:
The purpose of this cross-sectional, observational study is to evaluate the site and mechanism(s) for expiratory airflow limitation in chronic, treated, current or former smokers (>15 pack years) with COPD, Emphysema, and Asthma-COPD Overlap with mild to severe expiratory airflow limitation. Treatment may include short and long acting inhaled beta2agonists, short and long acting inhaled muscarinic receptor antagonists, inhaled and or oral corticosteroid, oral antibiotic, supplemental oxygen, and PDE type 4 inhibitor. In some cases, the patient may have had a history of asthma preceding the development of COPD (Asthma COPD Overlap).

DETAILED DESCRIPTION:
The investigators are interested in determining the predominant site of expiratory airflow limitation including large central airways vs small peripheral airways/alveoli. In mild to moderate obstructive airways disease and emphysema, I believe routine spirometry including FEV 1(L), FVC (L), and FEV 1/FVC % may be normal, despite expiratory airflow limitation in lung peripheral airways. I also want to determine whether the mechanism(s) of expiratory airflow limitation are related to measured loss of lung elastic recoil or intrinsic obstruction of small peripheral airways or both. It is also important to determine the extent and distribution of emphysema using high resolution, thin section lung CT with voxel quantification. If available pathological analysis of lung surgical specimens and also formalin inflated lungs obtained at autopsy will also be studied. Blood studies will include but not limited to CBC, serum IgE, complete metabolic panel, and alpha 1 antitrypsin levels. Extensive lung function testing will also include spirometry tests before and after inhaled albuterol bronchodilation, lung volumes measured in a plethysmograph, diffusing capacity, measurement of lung elasticity that requires placement of an esophageal balloon, measurement of airflow after breathing a mixture of 80% helium-20%oxygen for 7-10 minutes, and measurements of exhaled nitric oxide. CAT scans of the lungs will be obtained to evaluate the presence, extent and distribution of emphysema and bronchiectasis. In some cases, bronchoscopy may be requested.

The above tests may be uncomfortable but should cause no harm.

ELIGIBILITY:
Inclusion Criteria:

* asthma- copd overlap
* emphysema in smokers with smoking history > 15 pack years
* COPD/ bronchitis and bronchiectasis in smokers with smoking history
* >15 pack years

Exclusion Criteria:other pulmonary or systemic diagnosis

* non smokers
* any other pulmonary diagnosis
* pulmonary fibrosis

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Site and Mechanism(s) of Expiratory Airflow Limitation | 4 years
  Contribution of loss of lung lastic recoil vs intrinsic airway obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Arthur F Gelb, MD, Principal Investigator — Clin Prof Geffen School of Medicine at UCLA Medical Center; Arthur F Gelb, MD, Study Director — Clin Prof Geffen School of Medicine at UCLA Medical Center
Locations (1):
- Arthur F Gelb MD, Lakewood, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of tests
Supporting Information: Study Protocol, CSR
Time Frame: As indicated for collaborration
Access Criteria: within 2 weeks of testing

REFERENCES:
- [Result] Qaseem A, Wilt TJ, Weinberger SE, Hanania NA, Criner G, van der Molen T, Marciniuk DD, Denberg T, Schunemann H, Wedzicha W, MacDonald R, Shekelle P; American College of Physicians; American College of Chest Physicians; American Thoracic Society; European Respiratory Society. Diagnosis and management of stable chronic obstructive pulmonary disease: a clinical practice guideline update from the American College of Physicians, American College of Chest Physicians, American Thoracic Society, and European Respiratory Society. Ann Intern Med. 2011 Aug 2;155(3):179-91. doi: 10.7326/0003-4819-155-3-201108020-00008. PMID 21810710
- [Result] Alcaide AB, Sanchez-Salcedo P, Bastarrika G, Campo A, Berto J, Ocon MD, Fernandez-Montero A, Celli BR, Zulueta JJ, de-Torres JP. Clinical Features of Smokers With Radiological Emphysema But Without Airway Limitation. Chest. 2017 Feb;151(2):358-365. doi: 10.1016/j.chest.2016.10.044. Epub 2016 Nov 3. PMID 27818328
- [Result] Mannino DM, Make BJ. Is it time to move beyond the "O" in early COPD? Eur Respir J. 2015 Dec;46(6):1535-7. doi: 10.1183/13993003.01436-2015. No abstract available. PMID 26621878
- [Result] Rennard SI, Drummond MB. Early chronic obstructive pulmonary disease: definition, assessment, and prevention. Lancet. 2015 May 2;385(9979):1778-1788. doi: 10.1016/S0140-6736(15)60647-X. PMID 25943942
- [Result] Harvey BG, Strulovici-Barel Y, Kaner RJ, Sanders A, Vincent TL, Mezey JG, Crystal RG. Risk of COPD with obstruction in active smokers with normal spirometry and reduced diffusion capacity. Eur Respir J. 2015 Dec;46(6):1589-1597. doi: 10.1183/13993003.02377-2014. Epub 2015 Nov 5. PMID 26541521
- [Result] Johns DP, Walters JA, Walters EH. Diagnosis and early detection of COPD using spirometry. J Thorac Dis. 2014 Nov;6(11):1557-69. doi: 10.3978/j.issn.2072-1439.2014.08.18. PMID 25478197
- [Result] Woodruff PG, Barr RG, Bleecker E, Christenson SA, Couper D, Curtis JL, Gouskova NA, Hansel NN, Hoffman EA, Kanner RE, Kleerup E, Lazarus SC, Martinez FJ, Paine R 3rd, Rennard S, Tashkin DP, Han MK; SPIROMICS Research Group. Clinical Significance of Symptoms in Smokers with Preserved Pulmonary Function. N Engl J Med. 2016 May 12;374(19):1811-21. doi: 10.1056/NEJMoa1505971. PMID 27168432
- [Result] Rodriguez-Roisin R, Han MK, Vestbo J, Wedzicha JA, Woodruff PG, Martinez FJ. Chronic Respiratory Symptoms with Normal Spirometry. A Reliable Clinical Entity? Am J Respir Crit Care Med. 2017 Jan 1;195(1):17-22. doi: 10.1164/rccm.201607-1376PP. No abstract available. PMID 27598473
- [Result] Martinez CH, Diaz AA, Meldrum C, Curtis JL, Cooper CB, Pirozzi C, Kanner RE, Paine R 3rd, Woodruff PG, Bleecker ER, Hansel NN, Barr RG, Marchetti N, Criner GJ, Kazerooni EA, Hoffman EA, Ross BD, Galban CJ, Cigolle CT, Martinez FJ, Han MK; SPIROMICS Investigators. Age and Small Airway Imaging Abnormalities in Subjects with and without Airflow Obstruction in SPIROMICS. Am J Respir Crit Care Med. 2017 Feb 15;195(4):464-472. doi: 10.1164/rccm.201604-0871OC. PMID 27564413
- [Result] Regan EA, Lynch DA, Curran-Everett D, Curtis JL, Austin JH, Grenier PA, Kauczor HU, Bailey WC, DeMeo DL, Casaburi RH, Friedman P, Van Beek EJ, Hokanson JE, Bowler RP, Beaty TH, Washko GR, Han MK, Kim V, Kim SS, Yagihashi K, Washington L, McEvoy CE, Tanner C, Mannino DM, Make BJ, Silverman EK, Crapo JD; Genetic Epidemiology of COPD (COPDGene) Investigators. Clinical and Radiologic Disease in Smokers With Normal Spirometry. JAMA Intern Med. 2015 Sep;175(9):1539-49. doi: 10.1001/jamainternmed.2015.2735. PMID 26098755
- [Result] Gelb AF, Hogg JC, Muller NL, Schein MJ, Kuei J, Tashkin DP, Epstein JD, Kollin J, Green RH, Zamel N, Elliott WM, Hadjiaghai L. Contribution of emphysema and small airways in COPD. Chest. 1996 Feb;109(2):353-9. doi: 10.1378/chest.109.2.353. PMID 8620705
- [Result] Gelb AF, Schein M, Kuei J, Tashkin DP, Muller NL, Hogg JC, Epstein JD, Zamel N. Limited contribution of emphysema in advanced chronic obstructive pulmonary disease. Am Rev Respir Dis. 1993 May;147(5):1157-61. doi: 10.1164/ajrccm/147.5.1157. PMID 8484625
- [Result] Gelb AF, Yamamoto A, Verbeken EK, Nadel JA. Unraveling the Pathophysiology of the Asthma-COPD Overlap Syndrome: Unsuspected Mild Centrilobular Emphysema Is Responsible for Loss of Lung Elastic Recoil in Never Smokers With Asthma With Persistent Expiratory Airflow Limitation. Chest. 2015 Aug;148(2):313-320. doi: 10.1378/chest.14-2483. PMID 25950858
- [Result] Gelb AF, Gold WM, Wright RR, Bruch HR, Nadel JA. Physiologic diagnosis of subclinical emphysema. Am Rev Respir Dis. 1973 Jan;107(1):50-63. doi: 10.1164/arrd.1973.107.1.50. No abstract available. PMID 4683321
- [Result] Gelb AF, Zamel N. Simplified diagnosis of small-airway obstruction. N Engl J Med. 1973 Feb 22;288(8):395-8. doi: 10.1056/NEJM197302222880805. No abstract available. PMID 4684043
- [Result] Gelb AF, Williams AJ, Zamel N. Spirometry. FEV1 vs FEF25-75 percent. Chest. 1983 Oct;84(4):473-4. doi: 10.1378/chest.84.4.473. No abstract available. PMID 6617285
- [Result] Gelb AF, Yamamoto A, Mauad T, Kollin J, Schein MJ, Nadel JA. Unsuspected mild emphysema in nonsmoking patients with chronic asthma with persistent airway obstruction. J Allergy Clin Immunol. 2014 Jan;133(1):263-5.e1-3. doi: 10.1016/j.jaci.2013.09.045. Epub 2013 Nov 28. No abstract available. PMID 24290280
- [Result] Gelb AF, Yamamoto A, Verbeken EK, Schein MJ, Moridzadeh R, Tran D, Fraser C, Barbers R, Elatre W, Koss MN, Glassy EF, Nadel JA. Further Studies of Unsuspected Emphysema in Nonsmoking Patients With Asthma With Persistent Expiratory Airflow Obstruction. Chest. 2018 Mar;153(3):618-629. doi: 10.1016/j.chest.2017.11.016. Epub 2017 Nov 29. PMID 29197547